CLINICAL TRIAL: NCT00813111
Title: A Phase 3, Multicenter, Randomized, Double-blind Parallel-group, Active-control Study to Evaluate the Safety and Efficacy of Local Administration of SKY0402 for Prolonged Postoperative Analgesia in Subjects Undergoing Bilateral, Cosmetic Sub-muscular Breast Augmentation
Brief Title: Phase 3 Study of Local Administration of SKY0402 for Postoperative Analgesia in Subject Undergoing Breast Augmentation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision, unrelated to safety
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SIMPLE Breast Augmentation 315
Record Dates: First submitted 2008-12-09; First posted 2008-12-22 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-11

CONDITIONS: Pain
Keywords: Postsurgical pain; Analgesia; Breast augmentation
MeSH Terms: conditions — Pain; Pain, Postoperative; Agnosia | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKY0402 (Experimental): A single local administration of 300 mg in a 20-mL volume into each breast implant pocket for a total dose of 600 mg (i.e., a total of 40 mL)
  Interventions: Drug: SKY0402
- Bupivacaine HCl (Active Comparator): A single local administration of 100 mg in a 20-mL volume into each breast implant pocket for a total dose of 200 mg (i.e., a total of 40 mL)
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: SKY0402 — 600mg SKY0402 instilled into breast pocket during surgery
  Other Names: EXPAREL
  Arms: SKY0402
Drug: Bupivacaine HCl — 200mg Bupivacaine HCl instilled into breast pocket during surgery
  Other Names: Marcaine 0.5% with epinephrine
  Arms: Bupivacaine HCl

SUMMARY:
The purpose of this study is to provide a more effective postoperative method of pain control for patients undergoing cosmetic sub-muscular breast augmentation. Appropriate postoperative pain management contributes to faster patient mobilization, shortened hospital stays, and reduced healthcare costs.

DETAILED DESCRIPTION:
This is a phase 3 study conducted to evaluate the safety and efficacy of a single local administration of 300 mg of SKY0402 compared with 100 mg of conventional, commercially-available bupivacaine HCl (i.e. Marcaine 0.5% with epinephrine) administered locally into the implant pocket of each breast for postoperative analgesia in subjects undergoing bilateral, cosmetic, sub-muscular, breast augmentation under general anesthesia (endotracheal or otherwise). A total of 600 mg of SKY0402 or 200 mg bupivacaine HCl per subject is therefore administered. Post-operative assessments were conducted including adverse event and serious adverse event monitoring through Day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Women greater than or equal to 18 years of age at Screening Visit
2. Postmenopausal, surgically sterile, or willing to use acceptable means of contraception for at least 30 days after surgery including any of the following: hormonal contraceptives (e.g., oral, injectable, implantable starting at least 30 days before study administration), effective double-barrier methods (e.g., condoms with spermicide), intrauterine device, lifestyle with a personal choice of abstinence, nonheterosexual lifestyle, or a strictly monogamous relationship with a partner who has had a vasectomy.
3. Scheduled to undergo primary, bilateral, cosmetic, sub-muscular, breast augmentation under general anesthesia (endotracheal or otherwise)
4. American Society of Anesthesiologist (ASA) Physical Class 1-4
5. Able and willing to comply with all study visits and procedures, and with diary entries through postoperative day 8
6. Able to speak, read, and understand the language of the informed consent form (ICF), study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments
7. Willing and capable of providing written informed consent.

Exclusion Criteria:

A subject will not be eligible for the study if she meets any of the following criteria:

1. Women undergoing reconstructive surgery following mastectomy
2. Pregnancy, nursing, or planning to become pregnant during the study or within one month after study drug administration.
3. Use of any of the following medications within the times specified before surgery:

   1. long-acting opioids within 3 days.
   2. Any opioid medication within 24 hours.
4. Concurrent painful physical condition or concurrent surgery that may require analgesic treatment in the postoperative period for pain that is not strictly related to the surgical site being administered study drug (e.g., significant pain from other joints, chronic neuropathic pain, concurrent abdominal surgery, etc.), which have the potential to confound the postoperative study assessments.
5. Body weight less than 50 kilograms (110 pounds)
6. History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics, opioid medication, epinephrine, or sulfites.
7. Contraindication to epinephrine, such as concurrent administration of ergot-type drugs, monoamine oxidase (MAO) inhibitors or antidepressants of tryptoline or imipramine types, conditions where the production or exacerbation of tachycardia could provide fatal (e.g., poorly controlled thyrotoxicosis or severe heart disease) or any other pathological conditions that might be aggravated by the effect of epinephrine.
8. Administration of investigational product within 30 days of 5 elimination half-lives of such investigational product, whichever is longer, prior to study drug administration or planned administration of another investigational product or procedure during the subject's participation in this study.
9. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
10. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance with the protocol.
11. Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial, such as: debilitating diseases, acute illnesses, hypotension, partial or complete conduction block, impaired cardiac function, untreated hypertension, advanced arteriosclerotic heart disease, cerebral vascular insufficiency, pre-existing abnormal neurological or neuromuscular disease (e.g., epilepsy, myasthenia gravis), advanced liver disease, severe renal impairment, advanced diabetes, co-morbid conditions associated with an immunocompromised status such as blood dyscrasias, HIV/AIDS, or recent chemotherapy.

    In addition, the subject will be ineligible to receive study drug if she meets the following criteria during surgery:
12. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postoperative course.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Warnott, RN, Study Director — Pacira Pharmaceuticals, Inc
Locations (15):
- United States (15):
  - West Alabama Research, LLC., Birmingham, Alabama
  - West Alabama Research, LLC, Birmingham, Alabama
  - Horizon Research Group, Inc, Mobile, Alabama
  - La Jolla Spa MD, La Jolla, California
  - Associates for Plastic Surgery Medical Group, Inc., La Jolla, California
  - Lotus Clinical Research, Pasadena, California
  - Pacific Plastic Surgery, Santa Barbara, California
  - Miami Plastic Surgery, Miami, Florida
  - North Fulton Plastic Surgery, Roswell, Georgia
  - Waldman and Schantz Plastic Surgery, Lexington, Kentucky
  - Back Bay Plastic Surgery, Boston, Massachusetts
  - Personal Enhancement Center, Toms River, New Jersey
  - The Ohio State University Research Foundation, Columbus, Ohio
  - Research Concepts, Ltd, Bellaire, Texas
  - Office of Dr. William P. Adams, Jr., MD, University Park, Texas

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SKY0402 | Bupivacaine HCl
Started | 66 | 70
Completed | 64 | 70
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SKY0402 | Bupivacaine HCl | Total
Number analyzed (Participants) | 66 | 70 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 70 | 136
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (7.3) | 30.6 (7.6) | 30.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 70 | 136
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 70 | 136

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) With Activity (NRS-A) Pain Intensity Scores
Description: Assessments of postoperative pain included pain intensity at rest (using the NRS at rest [NRS-R] and with activity [using the NRS-A]) where the prescribed activity was raising both arms.
  Pain intensity was assessed on a scale of 0 to 10, where 0=no pain and 10=worst possible pain.
Time Frame: through 72 hours
Population: Note: 136 subjects were randomized and received study drug and were included in the analyses. 10 subjects were randomized but not dosed and 4 additional subjects failed screening, resulting in 122 subjects.
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Arm/Group | SKY0402 | Bupivacaine HCl
Number analyzed (Participants) | 60 | 62
Units on a scale*hours | 441 (163) | 467 (181)

2. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SKY0402 | Bupivacaine HCl
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/70
Other Adverse Events (participants affected / at risk) | 48/66 | 51/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SKY0402 (N=66) | Bupivacaine HCl (N=70)
nausea (Gastrointestinal disorders) | 29 | 37
vomiting (Gastrointestinal disorders) | 10 | 14
Constipation (Gastrointestinal disorders) | 11 | 13
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Chills (General disorders) | 4 | 2
Headache (Nervous system disorders) | 2 | 5
Hypoaesthesia (Nervous system disorders) | 4 | 3
Tachycardia (Cardiac disorders) | 3 | 7
Insomnia (Psychiatric disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No